CLINICAL TRIAL: NCT00559286
Title: Influence of the Angiotensin Receptor Blocker Telmisartan on the Red Blood Cell Function and the Microcirculatory Perfusion
Brief Title: Effect of the Known Antihypertensive Drug Telmisartan on Red Blood Cells and Circulation in the Smallest Blood Vessels
Acronym: ITEM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: logistic reasons, patients could not be recruited
Sponsor: RWTH Aachen University (Other)
Collaborators: CTCA (Unknown); Heidelberg University (Other); Bayer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AIX-MK-01; EUDRA CT No 2007-002765-12
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Arterial Hypertension; Diabetes Mellitus Type 2 IRC or NIR
Keywords: perfusion; microcirculation; RBC function; NO metabolism; AT receptor blocker
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): treatment with 80 mg Telmisartan per day for 30 days
  Interventions: Drug: Telmisartan
- B (Active Comparator): treatment with 20mg Telmisartan per day for 30 days
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Telmisartan — application of 80mg or 20mg Telmisartan per day for 30 days

SUMMARY:
The hypothesis of the presented study is: Telmisartan induces an increase of eNOS activity in RBC resulting in an enhanced intravascular NO bioavailability, an ameliorated RBC deformability and a reduction of RBC and platelet aggregation. This could be a potential mechanism of the improvement of microcirculatory disorders, especially in patients with diabetes mellitus and arterial hypertension, treated with Telmisartan.

DETAILED DESCRIPTION:
Recently, it could be shown that the renin-angiotensin-system (RAS) influences different signal transduction pathways within the red blood cells (RBC). This includes the Na+/H+ exchange activity, the Ca2+-ATP-ase mediated Ca2+efflux, the erythropoietin- dependent production of RBC, the RBC deformability, RBC aggregation and the interaction of RBC and platelets. Recent studies and experiments, done by our group, focus on the oxidative and nitrosative metabolism of NO within the blood. The interactions of the RAS and endothelial NO are well known and described in detail. Based on a wide experience in this research field of NO metabolism, we characterized recently an active endothelial-type NO-synthase in RBC on the biochemical, functional and molecular level. Erythrocyte-derived NO formation serves important regulatory functions essential for adequate passage of blood through the vasculature. Here we aimed to treat patients with diabetes mellitus and arterial hypertension with Telmisartan as an angiotensin receptor antagonist. Efficacy parameters studied in this study should be: i) RBC deformability, RBC aggregation, ii) RBC dependent production of nitric oxide as well as detection of eNOS activity in RBC and iii) indices of microcirculatory perfusion. This project could broaden the view of effects of Telmisartan in the treatment of microcirculatory disorders in patients with diabetes mellitus and arterial hypertension, who exhibit a reduced NO bioavailability and RBC function.

ELIGIBILITY:
Inclusion Criteria:

* Men older than 18 years
* Diabetes mellitus type 2 defined according to the criteria of the American Diabetes Association Arterial hypertension defined according to the criteria of the Joint National Committtees (JNC 7)
* Given informed consent

Exclusion Criteria:

* Serve heart failure
* Serve aortic valve stenosis or hypertrophy obstructive cardiomyopathy
* Relevant cardiac arrhythmias
* Acute myocardial infarction within the last 4 weeks
* renal failure
* bilateral renal artery stenosis
* liver diseases
* primary hyperaldosteronism
* orthostatic hypotension (systolic blood pressure <100mmHg)
* hypokalemia, hyponatremia, hypercalcemia, symptomatic hyperuricemia
* inflammatory disease
* malignant disease
* previous intolerance to AT1 receptor antagonists and/or sulfonamides
* current therapy with insulin sensitizer
* current therapy with digoxin
* known abuse of alcohol or drugs

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Changes in Elongation-Index (EI) Method: To determine the elongation index (EI) we use the Laser assisted optical rotational cell analyzer (Lorrca). | after 30 days of treatment with study drug/control

SECONDARY OUTCOMES:
Improvement of microcirculatory perfusion (using laser doppler measurement) | after 30 days treatment
Improvement of endothelial function (using ultrasound measurements during flow mediated dilation) | after 30 days treatment
Increase in the total blood born NO pool (using reductive gase phase chemiluminescence | after 30 days treatment
Decrease of RBC aggregation (using Laser assisted optical rotational cell analyzer (Lorrca) | after 30 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, MD, Univ.Prof., Principal Investigator — Department of Cardiology, Angiology, Pulmonary Diseases and cardiologic critical care
Locations (1):
- University Hospital, Aachen, North Rhine-Westphalia, Germany